CLINICAL TRIAL: NCT03082638
Title: Identification of Lipid Biomarkers of Inflammation and Metabolic Disturbances in Gulf War Illness (GWI)
Brief Title: Identification of Gulf War Illness (GWI) Biomarkers
Status: Completed | Type: Observational
Sponsor: Roskamp Institute Inc. (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: RI-GWI-001
Record Dates: First submitted 2017-03-13; First posted 2017-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2024-04

CONDITIONS: Gulf War Illness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be analyzed for lipids, proteins, DNA, RNA and breakdown products to identify biomarkers for GWI
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control: served in Gulf War during 1990 - 1991 and have no symptoms of Gulf War Illness based on criteria
- Case: Served in Gulf War during 1990 -1991 and have Gulf War Illness

SUMMARY:
The scientists working on this study want to use blood samples to identify components in blood, such as protein, lipids and their breakdown products to determine if they can be used for diagnosing Gulf War Illness (GWI). An additional goal is to examine the relationship of changes in these markers with the exposures and symptoms associated with GWI.

The Scientists will also prepare RNA and DNA from the blood samples for genetic analyses of certain proteins known to increase the risk for GWI. This information will be one of the factors included in the analysis of results from the protein studies.

DETAILED DESCRIPTION:
Research studies conducted over the last decade provide compelling evidence that Gulf War Illness (GWI) may have been caused by exposure to chemicals, such as an anti-nerve agent pyridostigmine bromide (PB) and different types of pesticides (GW agents). These studies also show that brain structures that are involved in processing and storing memory, as well as brain pathways involved in controlling pain and fatigue, are altered in GW veterans with this condition. Even now, nearly 25 years later, veterans with GWI continue to experience these complex symptoms and this illness remains difficult to diagnose since the current GWI diagnostic process are limited by having to use information on self-reporting of symptoms. As such, there remains a need for developing minimally invasive blood based disease markers (biomarker) of GWI. The goal of this current study is to identify novel biomarkers of GWI which can assist physicians in providing an objective diagnosis of GWI so that appropriate clinical evaluations and treatments can be provided to GW veterans with this condition. Another key goal of this project is to identify biomarkers of GW chemical exposure and symptom profiles so that care and treatment can be tailored individually for each veteran with GWI. Scientists working in the field of GWI research continue to provide strong evidence that this condition is connected with irregular responses by blood cells which generally combat irritations or other injuries to the body (inflammation). Scientists have also found that GWI could also be due to damage to mitochondria, known as the powerhouses responsible for generating energy through the breakdown of sugars and fats (lipids).

Scientists at the Roskamp Institute have developed mouse models of GWI in order to identify biomarkers of brain damage and neurobehavioral problems that are a direct consequence of chemicals to which GW veterans were exposed during the 1991 GW. They have identified that there might be problems with breaking down fats in the brains of exposed mice even long after subacute exposure to GW agents. In particular, they show changes in lipids which belong to cellular compartments (peroxisomes) that perform tasks similar to those of the mitochondria with respect to the breakdown of fats. The inflammatory processes, mitochondria and peroxisomes display unique lipid classes that can be measured in blood using mass spectrometry technologies. These technologies allow us to detect and measure elemental composition of each lipid. We plan to use this technology to study lipids that are specific to inflammation and metabolic disturbances associated with GWI in order to determine if they can be used as biomarkers of GWI. In collaboration with the Boston GWI consortium, we are testing this hypothesis and our early pilot work in control and GWI veterans support potential use of these lipids as biomarkers of GWI. The proposal will expand these pilot studies and determine if lipids associated with these key disturbances in GWI can be useful tools for diagnosing GWI. The proposal will also try to use these lipids in order to identify subgroups of GW veterans with similar chemical exposures and symptom patterns. This work will also be facilitated by the use of blood samples from GWI animal models that will help with translational studies linking animal model work and human studies. This will help fill the gaps between the two so that future studies can be conducted that can use these biomarkers to determine if treatments and care designed for GWI are succeeding.

Furthermore, identifying biomarkers of exposures and symptom profiles which will help with delivering personalized care and treatment to each veteran appropriately. The existing expertise and collaborations between the Roskamp Institute and the Boston GWI consortium will expedite successful translation of this endeavor so that appropriate biomarker tools are made available to the clinicians in order to assist them with diagnosing GWI and ensuring that appropriate medical plans are developed for the care and treatment of veterans with GWI.

ELIGIBILITY:
Inclusion Criteria:

1. Age 35 years or older 2. Served in the 1990-1991 Gulf War 3. Ability to understand written and spoken English or availability of a legal representative who can understand written or spoken English. Participants and caregiver/informants must be able to read, write and speak the language in which psychometric tests are provided with visual and auditory acuity (corrected) sufficient to allow for accurate testing.

-

Exclusion Criteria:

1. Diagnosed or being treated by a physician for any of the following (Steele et al, 2000) and deemed clinically significant per the discretion of the PI:
2. Cancer (except for non-melanoma skin cancers)
3. Chronic infectious disease
4. Problems resulting from postwar injuries.
5. Liver disease
6. Lupus
7. Multiple sclerosis
8. Stroke
9. Serious psychiatric condition (those associated with psychosis and/or for which the respondent had been hospitalized since 1991).
10. Hospitalized in the last 5 years for alcohol or drug dependence, depression, or post-traumatic stress disorder (PTSD).
11. Diagnosis of Dementia of any type or Parkinson's disease

    -

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Veterans who served in the Gulf War during 1990 to 1991
Sampling Method: Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Lipid bio markers | 2017 to 2019
  Determine if lipids specific to inflammation, mitochondria and peroxisome function can be objective biomarkers of the CNS pathology of GWI.

SECONDARY OUTCOMES:
Identification of Subgroups | 2017 to 2019
  determine if lipid biomarkers can identify subgroups of ill GW veterans based on symptom patterns and GW chemical exposures.

CONTACTS AND LOCATIONS:
Overall Officials: Laila Abdullah, PhD, Principal Investigator — The Roskamp Institute, Inc
Locations (1):
- The Roskamp Institute, Inc., Sarasota, Florida, United States

IPD SHARING:
Plan to Share IPD: No